CLINICAL TRIAL: NCT02504229
Title: DC-CIK In Combination With Chemotherapy ( Gio / Oxaliplatin or Cisplatin ) Versus First-line Chemotherapy for Locally Advanced Unresectable or Metastatic Gastric Adenocarcinoma Randomized Controlled Phase II Clinical Study of Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Biohealthcare Biotechnology Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC-A-004
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — gimeracil; Oxaliplatin

ARMS (2):
- Chemotherapy+DC-CIK (Experimental): Combined treatment group:mononuclear cells were obtained aseptically with blood cell separator composition spheresis 1 day before SOX program chemotherapy, cultured DC-CIK cells. SOX program was acted on Day 2. Cells were cultured 14d,2 times back to the patient.A 21d was a cycle, then evaluated the therapeutic effect after two cycles.
  Interventions: Biological: autologous dendritic cells co-cultured with cytokine-induced killer cells; Drug: Gimeracil and Oteracil Porassium Capsules; Drug: Oxaliplatin
- Chemotherapy alone (Active Comparator): Chemotherapy: two groups were treated with SOX program,specific drugs:Venoclysis of oxaliplatin 130mg/㎡;Day 1; Tegafur,Gimeracil and Oteracil Porassium Capsules 80mg/㎡/d,two oral/d;Day 1 to 12; 21d as one cycle of treatment, evaluated the therapeutic effect after two cycles.
  Interventions: Drug: Gimeracil and Oteracil Porassium Capsules; Drug: Oxaliplatin

INTERVENTIONS:
Biological: autologous dendritic cells co-cultured with cytokine-induced killer cells
  Arms: Chemotherapy+DC-CIK
Drug: Gimeracil and Oteracil Porassium Capsules
Drug: Oxaliplatin
  Other Names: Eloxatin

SUMMARY:
This study evaluates the therapeutic effects of autologous dendritic cells co-cultured with cytokine-induced killer cells (DC-CIK) combined with S-1 ((Tegafur, Gimeracil, and Oteracil Potassium) and oxaliplatin adjuvant chemotherapy in locally advanced unresectable or metastaticgastric cancer. Half of participants will receive DC-CIK combined with S-1 and oxaliplatin adjuvant chemotherapy,while the other half will receive S-1 and oxaliplatin adjuvant chemotherapy served as controls.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18y;
2. ECOG physical status 0-1;
3. The histologic diagnosis of stomach/gastroesophageal junction adenocarcinoma;
4. According to the RECIST 1.1 standard with measurable or evaluable lesion;
5. Accept swallow oral drug;
6. WBC≧4.0×10^9/L;ALC≧0.8×10^9/L;ANC≧1.5×10^9/L;PLT≧100×10^9/L;ALT,AST≦2.5 times of the normal limit;ALP≦2.5 times of the normal limit;TBIL﹤1.5 times of the normal limit;SCr﹤1 times of the normal limit;ALB≧30g/L;
7. The expected survival time of more than 3 months;
8. good compliance;
9. Provide written informed consent.

Exclusion Criteria:

1. Vital organs (heart,liver,kidney) function is serious dysfunction;
2. Patients received organ transplantation;
3. Patients with other malignant tumors or have occurred brain metastasis;
4. Patients with history of autoimmune disease;
5. Patients in pregnancy or breast-feeding period(women of child-bearing age need to check pregnancy test);
6. Patients with acute infection disease or in chronic active stage;
7. Patients with clear history of drug allergy or belong to allergic constitution;
8. Patients received chemotherapy,radiation therapy, immunosuppressive drugs (cyclosporine A,etc.) or other immune treatment in 4 weeks;
9. Patients received other clinical trials in 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-11; Primary Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: jinwan Wang, Principal Investigator — Chinese Academy of Medical Sciences Tumor Hospital; lin yang, Principal Investigator — Chinese Academy of Medical Sciences Tumor Hospital
Locations (1):
- Chinese Academy of Medical Sciences Tumor Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Ma X, Peng L, Wang J, Gao L, Zhang W, Lu X, Liu J, Yang L. Autologous CIK cells combined with chemotherapy as the first-line treatment for locally advanced or metastatic gastric cancer is safe and feasible. Front Immunol. 2023 Nov 1;14:1267369. doi: 10.3389/fimmu.2023.1267369. eCollection 2023. PMID 38022664